CLINICAL TRIAL: NCT03745612
Title: Effects of Time-Restricted Feeding on Weight Loss and Cardiometabolic Risk Factors in Obese Adults: a Randomized Clinical Trial
Brief Title: Time Restricted Feeding on Weight Loss and Cardio-protection (TREATY Trial)
Acronym: TREATY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NFEC-2018-145
Record Dates: First submitted 2018-11-15; First posted 2018-11-19 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Obesity; Time Restricted Feeding; Weight Loss; Calorie Restriction
MeSH Terms: conditions — Obesity; Intermittent Fasting; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRF (Experimental): Time restricted feeding
  Interventions: Behavioral: Time restricted feeding
- CER (Active Comparator): continuous energy restriction
  Interventions: Behavioral: Continuous Energy Restriction

INTERVENTIONS:
Behavioral: Time restricted feeding — Participants will receive a diet of 1500-1800kcal/d for men and 1200-1500kcal/d for women during a window of 8 h/d (8 am to 4 pm).
  Arms: TRF
Behavioral: Continuous Energy Restriction — Participants will follow receive a diet of 1500-1800kcal/d for men and 1200-1500kcal/d for women, without a restriction of feeding time.
  Arms: CER

SUMMARY:
Time restricted feeding (TRF) is a novel type of intermittent calorie restriction diet that involves eating a daily period of 8 hours or less. This is a randomized controlled trial to evaluate the effect of time restricted feeding (TRF) on weight loss and cardiometabolic risk factors in obese adults over 12 months compared to continuous energy restriction (CER).

ELIGIBILITY:
Inclusion Criteria:

1. Male of female aged between 18 and 75 years old;
2. Body mass index (BMI)of 28.0 to 45.0 kg/m2;

Exclusion Criteria:

1. History of HIV, hepatitis B or C (self-report) or active pulmonary tuberculosis;
2. Diagnosis of type 1 and type 2 diabetes;
3. History of malignant tumors;
4. Serious liver dysfunction or chronic kidney disease (AST or ALT > 3 times the upper limit of normal, or eGFR<30 ml/min/1.73 m2);
5. History of serious cardiovascular or cerebrovascular disease (angina, myocardial infarction or stroke) in the past 6 months;
6. History of severe gastrointestinal diseases or gastrointestinal surgery in the past 12 months;
7. History of Cushing's syndrome, hypothyroidism, acromegaly, hypothalamic obesity;
8. Being a smoker or having been a smoker in the 3 months prior to their screening visit;
9. Taking medications affecting weight or energy intake/energy expenditure in the last 6 months, including weight loss medications, antipsychotic drugs or other medications as determined by the study physician;
10. Currently participating in weight loss programs or weight change in the past 3 months (> 5% current body weight) ;
11. Women who are pregnant or plan to become pregnant;
12. Patients who cannot be followed for 24 months (due to a health situation or migration);
13. Patients who are unwilling or unable to give informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2021-07-24 (Actual); Study Completion 2021-07-28 (Actual)

PRIMARY OUTCOMES:
Change in body weight over 12 months | Baseline to 12 months

SECONDARY OUTCOMES:
Change in body composition | Baseline to 12 months
Change in waist circumference | Baseline to 12 months
Change in liver fat | Baseline to 12 months
Change in visceral fat | Baseline to 12 months
Change in HbA1c | Baseline to 12 months
Change in Blood pressure | Baseline to 12 months
Change in blood lipids | Baseline to 12 months
Change in insulin sensitivity | Baseline to 12 months
Change in β cell function | Baseline to 12 months
Change in pulse wave velocity (PWV) | Baseline to 12 months
Depression measured by the Patient Health Questionnaire-9 (PHQ-9) | Baseline to 12 months
Quality of sleep measured by the Pittsburgh sleep quality index (PSQI) | Baseline to 12 months
Quality of life measured by the 12-item Short-Form Health Survey Questionnaire (SF-12) | Baseline to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Huijie Zhang, MD,PhD, Principal Investigator — Department of Endocrinology and Metabolism, Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Liu D, Huang Y, Huang C, Yang S, Wei X, Zhang P, Guo D, Lin J, Xu B, Li C, He H, He J, Liu S, Shi L, Xue Y, Zhang H. Calorie Restriction with or without Time-Restricted Eating in Weight Loss. N Engl J Med. 2022 Apr 21;386(16):1495-1504. doi: 10.1056/NEJMoa2114833. PMID 35443107